CLINICAL TRIAL: NCT00210184
Title: Multicentric Phase II Trial: Evaluation of Efficacy and Safety of FOLFIRI Association Treatment in Patients 70 Years Old and More Presenting Gastric Cancer Locally Advanced or Metastatic
Brief Title: Evaluation of Efficacy and Safety of FOLFIRI Association Treatment in Patients 70 Years of Age and Older With Gastric Cancer
Acronym: CEPAFIRI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Bergonié (Other)
Collaborators: Novartis (Industry); Sanofi-Synthelabo (Industry); Aventis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IB2004-18; CEPAFIRI
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2021-09-16 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Gastric Cancer
Keywords: Chemotherapy; gastric cancer; geriatric evaluation; efficacy; safety
MeSH Terms: conditions — Stomach Neoplasms | interventions — Leucovorin

ARMS (1):
- Irinotecan associated to fluorouracil and leucovorin (Experimental): On D1, as a single 90-minute intravenous infusion diluted in 250 ml of saline (sodium chloride a 9 ‰), or isotonic glucose, at a dose of 180 mg/m2. Dosage adjustments are provided in case of severe toxicity.
  Then 5FU/ folinic acid: 400 mg/m2 of 5-FU as an IV bolus followed by a continuous 2400 mg/m2 infusion over 46 hours with 400 mg/m2 of folinic acid or 200 mg/m2 of l-folinic acid as a 2-hour infusion before 5-FU administration.
  Doses of 5-FU are adjusted according to clinical tolerance. Resume on D15 for 6 months
  Interventions: Drug: Irinotecan associated to fluorouracil and leucovorin

INTERVENTIONS:
Drug: Irinotecan associated to fluorouracil and leucovorin

SUMMARY:
The number of patients over 70 years old with cancer is increasing in France. This population is heterogenous: physiological functions, presence of co-morbidities, and autonomy can vary a lot between subjects of the same age. Physicians hesitate to treat them with optimal doses because they are afraid of the risk of toxicity in spite of the benefits of treatment. Fifty eight percent of gastric cancers are diagnosed in patients over the age of 70 in France. FOLFIRI (irinotecan, leucovorin and fluorouracil) chemotherapy appears to be a promising treatment for digestive cancer. It increases the level of response and survival without major toxicity. It becomes necessary to evaluate patients, to propose adapted treatments for their conditions.

The principal objectives are to demonstrate the efficacy of treatment, safety, survival and to find out if geriatric assessment data can help to better predict chemotherapy toxicity. The researchers plan to accrue 43 patients diagnosed with locally advanced or metastatic gastric cancer. They will receive FOLFIRI and 4 geriatric evaluations: before treatment, day 1 cycle 2, day 1 cycle 4 and at the end of chemotherapy. These evaluations include tests of cognitive functions (MMS), nutritional status (MNA), co-morbidity (CIRS-G), mobility (Get up and Go), activities (ADL; IADL), quality of life (QLQ-C30), depression (GDS-15) and Lachs-Balducci screening.

ELIGIBILITY:
Inclusion Criteria:

* 70 years of age or older
* Gastric cancer, locally advanced or metastatic
* No previous adjuvant treatment (surgery, radiotherapy, chemotherapy) in the last 6 months
* One measurable lesion
* ECOG < 3
* Biology and biochemistry within normal limits
* Life expectancy > 12 weeks

Exclusion Criteria:

* Other palliative chemotherapy for this cancer
* Other cancer in the last 5 years
* Previous treatment with irinotecan
* Atropine treatment not possible
* Concomitant cancer therapy except bone radiotherapy
* Metastases to brain or meninges with symptoms
* Other severe pathology uncontrolled
* Problem of compliance

Ages: 70 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 42 (Actual)
Dates: Start 2004-07-21 (Actual); Primary Completion 2009-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marianne FONCK, MD, Principal Investigator — Institut Bergonié
Locations (6):
- France (6):
  - Centre Hospitalier Universitaire de Bordeaux, Bordeaux
  - Institut Bergonié - Centre Régional de Luttre Contre le Cancer de Bordeaux et du Sud Ouest, Bordeaux
  - Hopital Robert Boulin, Libourne
  - Centre Hospitalier Universitaire de Pau, Pau
  - Clinique Francheville, Périgueux
  - Centre Hospitalier Universitaire de Villeneuve sur Lot, Villeneuve-sur-Lot

REFERENCES:
- [Result] Fonck M, Brunet R, Becouarn Y, Legoux JL, Dauba J, Cany L, Smith D, Auby D, Terrebonne E, Traissac L, Mertens C, Soubeyran P, Bellera C, Rainfray M, Mathoulin-Pelissier S. Evaluation of efficacy and safety of FOLFIRI for elderly patients with gastric cancer: a first-line phase II study. Clin Res Hepatol Gastroenterol. 2011 Dec;35(12):823-30. doi: 10.1016/j.clinre.2011.08.002. Epub 2011 Sep 8. PMID 21907007

RESULTS

PARTICIPANT FLOW:
Groups:
- Irinotecan Associated to Fluorouracil and Leucovorin: On D1, as a single 90-minute intravenous infusion diluted in 250 ml of saline (sodium chloride a 9 ‰), or isotonic glucose, at a dose of 180 mg/m2. Dosage adjustments are provided in case of severe toxicity.
  Then 5FU/ folinic acid: 400 mg/m2 of 5-FU as an IV bolus followed by a continuous 2400 mg/m2 infusion over 46 hours with 400 mg/m2 of folinic acid or 200 mg/m2 of l-folinic acid as a 2-hour infusion before 5-FU administration.Doses of 5-FU are adjusted according to clinical tolerance. Resume on D15 for 6 months.
Period: Overall Study
Arm/Group | Irinotecan Associated to Fluorouracil and Leucovorin
Started | 42
Completed | 40
Not Completed | 2
Not completed — The medical record was lost for these patients: no clinical data is available | 2

BASELINE CHARACTERISTICS:
Groups:
- Irinotecan Associated to Fluorouracil and Leucovorin: On D1, as a single 90-minute intravenous infusion diluted in 250 ml of saline (sodium chloride a 9 ‰), or isotonic glucose, at a dose of 180 mg/m2. Dosage adjustments are provided in case of severe toxicity.
  Then 5FU/ folinic acid: 400 mg/m2 of 5-FU as an IV bolus followed by a continuous 2400 mg/m2 infusion over 46 hours with 400 mg/m2 of folinic acid or 200 mg/m2 of l-folinic acid as a 2-hour infusion before 5-FU administration.
  Doses of 5-FU are adjusted according to clinical tolerance. Resume on D15 for 6 months
  Translated with www.DeepL.com/Translator (free version)
  Irinotecan associated to fluorouracil and leucovorin
Arm/Group | Irinotecan Associated to Fluorouracil and Leucovorin
Number analyzed (Participants) | 42
Age, Continuous [Median (Full Range); unit: years] | 77.3 [70.4 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 31
Region of Enrollment [Count of Participants; unit: Participants]
  France | 42

OUTCOME MEASURES:

1. Primary Outcome: 2-month Response Rate
Description: Response rate is defined as the rate of participants with partial or complete responses according to RECIST V1.0.
  Complete response is defined as the disappearance of all target lesions and partial response is defined as at least a 30% decrease in the sum of the longest diameters (SLD) of target lesions, taking as reference the baseline SLD (RECIST V1.0.).
Time Frame: 2 months
Population: The medical record was lost for 2 patients: no radiologial and clinical data is available
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Irinotecan Associated to Fluorouracil and Leucovorin
Number analyzed (Participants) | 40
percentage of participants | 25 [12.7 to 41.2]

2. Secondary Outcome: Overall Survival
Description: OS was defined as the time from trial inclusion to death due to any cause. Participants without documented death were censored at the date of the last follow-up or last patient contact. The OS was calculated using the product-limit (Kaplan-Meier) method for censored data.
Time Frame: From date of inclusion until the date of date of death from any cause, assessed up to 12 months.
Population: The medical record was lost for 2 patients: no radiologial and clinical data is available.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Irinotecan Associated to Fluorouracil and Leucovorin
Number analyzed (Participants) | 40
months | 10 [7 to 15]

3. Secondary Outcome: Progression-free Survival
Description: PFS was defined as time since trial inclusion to progression or death from any cause, whichever occurred first, and data from patients progression-free and lost to follow-up before the study end were censored at date of last news. The PFS was calculated using the product-limit (Kaplan-Meier) method for censored data. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From date of inclusion until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
Population: The medical record was lost for 2 patients: no radiologial and clinical data is available.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Irinotecan Associated to Fluorouracil and Leucovorin
Number analyzed (Participants) | 40
months | 7 [5 to 10]

ADVERSE EVENTS:
Description: Only serious adverse events were monitored. Adverse events (non-serious) were not assessed/monitored during the study.
Arm/Group | Irinotecan Associated to Fluorouracil and Leucovorin
All-Cause Mortality (participants affected / at risk) | 35/41
Serious Adverse Events (participants affected / at risk) | 16/41
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Irinotecan Associated to Fluorouracil and Leucovorin (N=41)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 3 (5)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Perocarditis (Cardiac disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
General disorders and administration site conditions - other specify (General disorders) | 4 (4)
Device related infection (Infections and infestations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
vomiting (Gastrointestinal disorders) | 1 (1)
Peritoneal infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes